CLINICAL TRIAL: NCT06942897
Title: Pilot Study for the Evaluation of a Dietary Supplement Containing Melissa Officinalis Formulated in Phospholipids on Mood Well-being and Cortisol Modulation
Brief Title: Evaluation of a Dietary Supplement Containing Melissa Officinalis Formulated in Phospholipids on Mood Well-being and Cortisol Modulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1267/21092023
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Stress; Mood Disorders; Emotional Well-being
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melissa Officinalis Supplement (Experimental): Participants will receive a dietary supplement containing 400 mg of Melissa officinalis formulated in phospholipids once daily for 3 weeks.
  Interventions: Dietary Supplement: Melissa officinalis supplement

INTERVENTIONS:
Dietary Supplement: Melissa officinalis supplement — This intervention consists of a standardized oral dietary supplement containing 400 mg of Melissa officinalis extract formulated in phospholipids. The supplement is administered once daily for 3 weeks to evaluate its potential effects on mood, stress perception, and cortisol levels in healthy adults.

SUMMARY:
This is a randomized, double-blind, placebo-controlled pilot study designed to evaluate the effect of an oral nutritional supplement containing Melissa officinalis formulated in phospholipids on mood and cortisol levels in healthy adults. Participants will be randomly assigned to receive either the active supplement or a placebo daily for 3 weeks. The primary outcome measures include changes in mood well-being, perceived stress, and salivary cortisol levels. The study aims to assess both efficacy and safety of the supplement in modulating stress response and emotional balance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Healthy volunteers as assessed by medical history and physical examination
* Willingness to comply with the study procedures

Exclusion Criteria:

* Current use of medications or supplements that may affect mood or cortisol levels
* Known allergy or sensitivity to Melissa officinalis or phospholipids
* History of psychiatric disorders (e.g., major depression, anxiety disorders)
* Significant comorbidities (e.g., cardiovascular, hepatic, renal diseases)
* Pregnant or breastfeeding women
* Participation in another clinical trial in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress levels measured by the Perceived Stress Scale (PSS) | week 4 (after 3 weeks of intervention)
  The PSS is a validated 10-item questionnaire that assesses the perception of stress over the past month. Scores range from 0 to 40, with higher scores indicating greater stress. The change from baseline to 3 weeks will be measured.